CLINICAL TRIAL: NCT06460142
Title: Multimodal Assessment of Biomarkers for Diagnosing Giant Cell Arteritis and Polymyalgia Rheumatica: A Comprehensive Analysis of Clinical, Laboratory, and Imaging Profiles
Brief Title: Assessing Biomarker in Giant Cell Arteritis and Polymyalgia Rheumatic
Acronym: GCAIO
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, Univ. Prof. Dr. med. Valentin Sebastian Schäfer, University Hospital, Bonn
Other Study IDs: 321/22
Record Dates: First submitted 2024-05-05; First posted 2024-06-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatica
Keywords: Giant Cell Arteritis; Polymyalgia Rheumatica; Vasculitis; Inflammatory Disorders; Clinical Biomarkers; Predictive Biomarkers; Disease Activity Monitoring; Therapeutic Response; Diagnostic Imaging Techniques; Aortic Imaging; Magnetic Resonance Imaging (MRI); Vascular Ultrasound; Optical Coherence Tomography Angiography (OCT-A); Transcriptome Analysis; Vascular-adhesion protein 1; Positron emission tomography-computed tomography (PET/CT); Siglec-9
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica; Vasculitis | interventions — Fluorescein Angiography; Optical Imaging; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC, Pax-Tube, Serum, Temporal artery biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PMR/ GCA: Patients diagnosed with GCA and/or PMR will be enrolled in this cohort. They will undergo a series of interventions including immunological profiling (cytokine profiling and immune cell phenotyping using flow cytometry, ELISA, 3'mRNA sequencing, high content analysis via a cell-based ex-vivo assay), and diagnostic imaging (MRI, OCTA including further ophthalmological assessment, vascular and transorbital ultrasound. Samples will be collected from patients at various stages of the disease (t=0, t=6, t=12, t=18 months, during flare-ups). Furthermore, TAB will be stained with a VAP-1 antibody to assess the expression and localization of VAP-1 in the arterial tissue.
  Interventions: Diagnostic Test: Aortic/ cardiac magnetic resonance imaging; Diagnostic Test: Vascular ultrasound; Diagnostic Test: Transorbital Ultrasound; Diagnostic Test: Contrast-Enhanced Ultrasound; Diagnostic Test: Optical coherence tomography angiography; Diagnostic Test: Fluorescein angiography; Diagnostic Test: Fundus autofluorescence; Diagnostic Test: Color Fundus Photography; Diagnostic Test: Cell-based ex-vivo assay with high-content analysis; Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay; Diagnostic Test: Flow cytometry; Diagnostic Test: Laboratory assessment:; Diagnostic Test: Immunohistochemistry of Temporal Artery Biopsies; Diagnostic Test: Functional assessment questionnaires
- Control Group: Age- and gender-matched healthy subjects will serve as the control group to provide baseline data for comparative purposes. This group will not receive any treatment related to GCA or PMR but undergoes similar diagnostic procedures for baseline measurements, including imaging and immunological assessments.
  Interventions: Diagnostic Test: Aortic/ cardiac magnetic resonance imaging; Diagnostic Test: Vascular ultrasound; Diagnostic Test: Transorbital Ultrasound; Diagnostic Test: Contrast-Enhanced Ultrasound; Diagnostic Test: Optical coherence tomography angiography; Diagnostic Test: Fluorescein angiography; Diagnostic Test: Fundus autofluorescence; Diagnostic Test: Color Fundus Photography; Diagnostic Test: Cell-based ex-vivo assay with high-content analysis; Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay; Diagnostic Test: Flow cytometry; Diagnostic Test: Laboratory assessment:; Diagnostic Test: Functional assessment questionnaires

INTERVENTIONS:
Diagnostic Test: Aortic/ cardiac magnetic resonance imaging — MRI scans will be performed to detect systemic vascular involvement in GCA patients, aiming to provide detailed images of affected tissues.
  Other Names: Aortic/ cardiac MRI
Diagnostic Test: Vascular ultrasound — Vascular ultrasound will be employed to examine the temporal and axillary arteries in GCA patients, searching for signs indicative of active inflammation.
Diagnostic Test: Transorbital Ultrasound — Transorbital ultrasound will be employed to assess the ophthalmic artery and its branches in GCA patients to detect intracranial inflammatory processes that could lead to severe neuro-ophthalmological complications.
  Other Names: TOS
Diagnostic Test: Contrast-Enhanced Ultrasound — Contrast-Enhanced Ultrasound (CEUS) is utilized to evaluate aortic involvement in GCA patients as an alternative, bed-side, realtime, radiation-free diagnostic tool.
  Other Names: CEUS
Diagnostic Test: Optical coherence tomography angiography — OCTA will be used to assess vascular changes in the retina of GCA patients, providing detailed imaging that can help detect early signs of ocular involvement and identify risk factors of anterior ischemic optic neuropathy.
  Other Names: OCTA
Diagnostic Test: Fluorescein angiography — Fluorescein angiography will be performed to evaluate blood circulation and highlight any blockages in the blood vessels of the retina in patients with GCA to detect vascular abnormalities that may lead to severe vision complications.
Diagnostic Test: Fundus autofluorescence — This imaging technique will be used to observe the health of the retina and detect any changes in GCA patients that could suggest disease activity, particularly useful for assessing the integrity of the retinal pigment epithelium.
Diagnostic Test: Color Fundus Photography — Color fundus photography will be used to document the appearance of the optic disc and retinal vasculature in GCA patients, aiding in the long-term monitoring of ocular changes and the effects of therapeutic interventions.
Diagnostic Test: Cell-based ex-vivo assay with high-content analysis — This assay predicts individual patient responses to different DMARDs by analyzing patient-derived PBMCs for specific immune responses to therapeutic agents.
  Other Names: GCAIO-essay
Diagnostic Test: 3'mRNA sequencing — 3'mRNA sequencing analyzes gene expression profiles related to the immune response in PMR/GCA patients, aiding in understanding the genetic underpinnings of inflammation and vascular remodeling.
Diagnostic Test: Enzyme-linked immunosorbent assay — Used to measure cytokine levels in the serum and plasma of PMR/GCA patients, ELISA aids in profiling inflammatory markers that are indicative of disease activity and response to treatment.
  Other Names: ELISA
Diagnostic Test: Flow cytometry — Employed to analyze immune cell phenotypes in patients with PMR and/or GCA, this test helps identify various immune cell subsets and their activation states, which are critical for understanding disease mechanisms and guiding therapy.
  Other Names: FACS
Diagnostic Test: Laboratory assessment: — Serum Chemistry (nt-proBNP, troponin T, CRP, ESR, blood count)
Diagnostic Test: Immunohistochemistry of Temporal Artery Biopsies — Immunohistochemistry staining of TAB to assess local expression of endothelial adhesion molecules in acute inflammation.
  Other Names: IHC TAB
  Groups: PMR/ GCA
Diagnostic Test: Functional assessment questionnaires — The following questionnaires will be applied: FACIT-Fatigue, SF-36, BAS, Birmingham Vasculitis Activity Score, Montreal Cognitive Assessment, Mini-Mental Status Examination. These questionnaires collectively provide a comprehensive evaluation of the functional status, quality of life, and mental health of patients with GCA and PMR.

SUMMARY:
The GCAIO study is an innovative, multimodal research initiative designed to enhance the understanding, diagnosis, and management of giant cell arteritis (GCA) and frequently associated polymyalgia rheumatica (PMR). This longitudinal study aims to dissect the complex immunological landscape and systemic manifestations of these conditions through a combination of diagnostic imaging and detailed immunological profiling.

The study focuses on three primary objectives: (1) Identifying and analyzing cytokine profiles and immune cell phenotypes, employing techniques like flow cytometry, enzyme-linked immunosorbent assays (ELISA), and next-generation sequencing to predict disease activity and therapeutic responses. (2) Advancing diagnostic and monitoring capabilities through the application of novel and established imaging technologies, including MRI, optical coherence tomography angiography (OCTA), and ultrasound. These modalities aim to improve the detection of neuro-ophthalmological, cardiac, and aortic complications in GCA, potentially offering more precise monitoring and earlier diagnosis. (3) Enhancing the understanding of PMR within the context of GCA by exploring specific biomarkers and advanced imaging to refine diagnostic accuracy and treatment strategies, thus improving patient outcomes.

DETAILED DESCRIPTION:
GCA is an immune-mediated vasculitis that affects medium and large-sized vessels, leading to vascular changes and occlusion due to severe vascular inflammation, neoangiogenesis, and remodeling. GCA has the potential to impact almost any organ. Despite advancements in understanding the pathophysiology and clinical manifestations of GCA, many aspects of the disease remain unexplored. The GCAIO study aims to fill these gaps using an integrative research approach to enhance the diagnosis, understanding, and management of GCA.

The GCAIO study cohort includes patients at their first diagnosis, throughout the disease, and during recurrent activity, facilitating a thorough longitudinal analysis of GCA. The research focuses on the complex immunological processes of the disease. Techniques such as flow cytometry (FACS), enzyme-linked immunosorbent assays (ELISA), and 3'-mRNA transcriptome analysis are employed to identify biomarkers that can assess GCA activity, track disease progression, and predict therapeutic responses, particularly for those unresponsive to interleukin (IL)-6 receptor (R) inhibitors. Additionally, the project is pioneering personalized treatment protocols tailored to individual immune profiles by developing a cell-based ex-vivo assay designed to forecast how patients will respond to different disease-modifying anti-rheumatic drugs (DMARDs).

Alongside the immunological research, the project emphasizes improving diagnostic and monitoring techniques through imaging technologies. Recent advancements have demonstrated that optimized diagnostics significantly enhance treatment outcomes for GCA patients. The planned prospective multimodal imaging aims to investigate potential neuro-ophthalmological, cardiac, and aortic manifestations during the course of GCA, enabling a detailed assessment of the involvement of various structures. Established imaging methods such as magnetic resonance imaging (MRI), optical coherence tomography angiography (OCTA), and vascular ultrasound are being extended into new areas to evaluate their diagnostic and prognostic merits. Furthermore, the investigators are exploring innovative diagnostic tools like transorbital ultrasound (TOS) and contrast-enhanced ultrasound (CEUS) for their potential as predictive biomarkers, facilitating earlier diagnosis and more precise disease monitoring. By correlating imaging findings with immunological data, our goal is to alter the way GCA is detected and monitored.

The inclusion of patients with PMR enhances our understanding of its pathophysiology, clinical manifestations, and its connection to often-associated GCA. The investigators are dedicated to developing new diagnostic criteria and exploring alternative therapeutic approaches for PMR maintenance therapy. By identifying alternative clinical, laboratory, or instrumental diagnostic methods to predict PMR, the investigators aim to set new diagnostic standards and deepen our understanding of its pathophysiology and immunological processes.

In summary, the goal of the GCAIO study is to make substantial contributions to the fields of GCA and PMR by developing innovative diagnostic and therapeutic strategies that improve treatment and quality of life for affected patients. The identification of specific biomarkers and the establishment of new diagnostic standards could lead to more precise diagnoses and optimized management of therapy, thereby enhancing patient care and reducing the risk of complications and therapy failures.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Participants (>18 years) must provide written informed consent to voluntarily participate in the study.
* Confirmed Diagnosis: Diagnosis of GCA or PMR confirmed by the treating physician and fulfilling expanded ACR-EULAR classification criteria. Patients must have been either newly diagnosed within the last three days or have experienced a disease flare within the same timeframe.

Exclusion Criteria:

* Severe Renal Insufficiency: Chronic glomerular filtration rate (GFR) less than 30 mL/min.
* Other Medical Conditions Requiring Glucocorticoids: Presence of medical conditions other than GCA or PMR that necessitate continuous or intermittent treatment with oral or parenteral glucocorticoids.
* Other Inflammatory Rheumatic Diseases: Patients with other inflammatory rheumatic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The GCAIO study focuses on patients with newly diagnosed GCA and PMR or those experiencing a flare-up. The primary sites for patient recruitment include the ophthalmological and rheumatological departments of the University Hospital of Bonn, Germany. Additional participants can be referred by local rheumatologists and primary care physicians. Healthy controls are recruited through the ophthalmological and rheumatological department of the University Hospital Bonn.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Detected Neuro-Ophthalmological Manifestations | At baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Use of OCTA, TOS, and additional ocular imaging to assess and monitor ocular and cranial vascular abnormalities indicative of GCA. Unit of Measure: Number of participants.
Number of Participants with Detected Cardiac and Aortic Involvement | At baseline, 6 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Detection and monitoring of inflammatory changes and structural anomalies in the cardiac and aortic regions using MRI and CEUS. Unit of Measure: Number of participants.
Changes in Immune Cell Phenotype | At baseline, 6 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Identification and quantification of immune cell types including changes over time using FACS. Unit of Measure: Changes in levels (percentages).
Changes in Cytokine Profiles | At baseline, 6 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Identification and quantification of cytokines including changes over time using 3'-mRNA transcriptome analysis. Unit of Measure: Changes in levels (pg/mL).
Levels of Siglec-9 in Blood | At baseline, 6 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Measurement of Siglec-9 levels on immune cells including changes over time using FACS. Correlation with clinical assessments of disease activity and imaging findings. Unit of Measure: Changes in levels (percentages).
Levels of sVAP-1 in Blood | At baseline, 6 months, 12 months, 18 months, and during flare-ups (assessed up to 18 months after diagnosis).
  Measurement of sVAP-1 levels in blood via ELISA including changes over time. Correlation with clinical assessments of disease activity and imaging findings. Unit of Measure: Changes in levels (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Valentin S. Schäfer, Univ. Prof., Principal Investigator — Department of Rheumatology and Clinical Immunology, University Hospital Bonn
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data are available upon reasonable request from the corresponding investigator.

REFERENCES:
- See also: Vasculitis Research Group Bonn (VAREGBO) — http://www.ukbonn.de/rheumatologie/unsere-forschung/varegbo/